CLINICAL TRIAL: NCT06854367
Title: Accelerated vs. Conventional Theta Burst Stimulation for Late-life Depression
Acronym: ACT-LLD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CTO4933
Record Dates: First submitted 2025-02-21; First posted 2025-03-03 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-02

CONDITIONS: Late Life Depression (LLD); Depression - Major Depressive Disorder; Depressive Disorder, Treatment-Resistant; Mood Disorders
Keywords: Brain stimulation; rTMS; Theta burst stimulation; Accelerated theta burst stimulation
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Mood Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Accelerated TBS (Active Comparator): Multiple treatments a day (5 treatments/day) for 4 consecutive days in the first week and 2 non-consecutive days in the second week.
  Interventions: Device: TBS
- Conventional TBS (Active Comparator): Treatment once a day for 30 days (e.g., 5 days a week for 6 weeks)
  Interventions: Device: TBS

INTERVENTIONS:
Device: TBS — Repetitive transcranial magnetic stimulation (rTMS) is a form of non-invasive neurostimulation that uses focused magnetic field pulses to directly stimulate cortical neurons. Theta burst stimulation (TBS) is a briefer form of patterned rTMS that has been shown to be effective against major depressive disorder. Each treatment will consist of either 1) cTBS of right DLPFC followed by iTBS of left DLPFC; or 2) iTBS of left DLPFC.

SUMMARY:
The purpose of this trial is to compare the treatment efficacy (improvement in depressive symptoms) of accelerated TBS protocol (where participants receive multiple TBS treatments daily) to conventional TBS protocol (where participants receive a single TBS treatment daily) in late life depression. In addition, the study also aims to determine if specific patterns of stimulation are more or less effective. To do this, all participants will receive active treatments, but some of the participants in this study will receive accelerated TBS and some will receive once daily TBS.

DETAILED DESCRIPTION:
The purpose of this trial is to compare the treatment efficacy (change in MADRS scores) of accelerated TBS to conventional TBS in participants with moderate to severe LLD at 4-weeks following accelerated TBS or following 30 once daily treatments of conventional TBS. Accelerated TBS group will receive 5 treatment sessions per day at approximately 1 hour intervals for 4 consecutive days on week 1 and 2 non-consecutive days on week 2. Conventional TBS group will receive 30 once daily treatment (approximately 6 weeks). Each treatment will consist of either 1) cTBS of right DLPFC followed by iTBS of left DLPFC; or 2) iTBS of left DLPFC.

ELIGIBILITY:
Inclusion Criteria:

1. are voluntary and competent to consent to treatment
2. are an outpatient
3. are ≥ 60 years old
4. have a Mini International Neuropsychiatric Interview (MINI 7.0) confirmed diagnosis of MDD, with a current MDE
5. have failed to achieve a clinical response to an adequate dose of an antidepressant based on an Antidepressant Treatment History Form (ATHF) score of ≥ 3 in the current episode or have failed to tolerate two separate trials of an antidepressant
6. have a score ≥ 10 on the Patient Health Questionnaire (PHQ-9)
7. have had no increase or initiation of any antidepressant or antipsychotic medication in the 4 weeks prior to screening
8. are able to adhere to the treatment schedule
9. pass the TMS adult safety screening (TASS) questionnaire

Exclusion Criteria:

1. have a Mini International Neuropsychiatric Interview (MINI 7.0) confirmed diagnosis of substance dependence or abuse within the last 3 months
2. have a concomitant major unstable medical illness as determined by one of the study physicians
3. have active suicidal intent
4. have presumed or probable dementia or clinical evidence of dementia as assessed by Short Blessed Test score ≥ 10
5. have a lifetime MINI diagnosis of bipolar I or II disorder, or primary psychotic disorder
6. have current psychotic symptoms
7. have a diagnosis of obsessive compulsive disorder, post-traumatic stress disorder (current or within the last year), anxiety disorder (generalized anxiety disorder, social anxiety disorder, panic disorder), or dysthymia, assessed by a study investigator to be primary and causing greater impairment than MDD
8. have a diagnosis of any personality disorder as assessed by a study investigator to be primary and causing greater impairment than MDD
9. did not respond to a course of ECT in the current depressive episode
10. have received rTMS in the current episode; patients who have had rTMS in a previous episode would be eligible
11. have a history of a primary seizure disorder or a seizure associated with an intracranial lesion
12. have an intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed
13. have an implanted electronic device that is currently in function such as a defibrillator
14. have a non-correctable clinically significant sensory impairment (i.e., cannot hear well enough to cooperate with interview)
15. have clinically significant laboratory abnormality, in the opinion of a study investigator
16. currently take more than lorazepam 2 mg daily (or equivalent) or any dose of an anticonvulsant
17. if participating in psychotherapy, must have been in stable treatment for at least 3 months prior to entry into the study, with no anticipation of change in the frequency of therapeutic sessions, or the therapeutic focus over the duration of the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2029-11 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Depression severity | 6 weeks
  Montgomery Asberg Depression Rating Scale (MADRS) Change

SECONDARY OUTCOMES:
Depression severity | up to 10 weeks
  17 item Hamilton Depression Rating Scale (HDRS-17) Change
Depression severity | up to 10 weeks
  The Beck Depression Inventory (BDI-II) Change
Anxiety severity | up to 10 weeks
  General Anxiety Disorder-7 (GAD-7) Change
Suicidal ideation | up to 10 weeks
  The Beck Scale for Suicide Ideation (BSS) Change
Global cognition | up to 10 weeks
  Montreal Cognitive Assessment (MoCA) Change
Executive function | up to 10 weeks
  Delis-Kaplan Executive Function System (D-KEFS) Change
Executive function | up to 10 weeks
  NIH Toolbox Flanker Inhibitory Control and Attention Test
Memory | up to 10 weeks
  California Verbal Learning Test- third edition (CVLT-3) Change
Disability and Functional Impairment | up to 10 weeks
  Sheehan Disability Scale (SDS) Change
Quality of Life Measure | up to 10 weeks
  Quality of Life Enjoyment and Satisfaction Scale (Q-LES-Q) change
Quality of Life Measure | up to 10 weeks
  World Health Organization Quality of Life Short Version (WHOQOL-BREF) Change
Participant Expectancy of Improvement and Preference | Baseline
  Modified Stanford Expectations of Treatment Scale (SETS)

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Centre for Addiction and Mental Healh, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided